CLINICAL TRIAL: NCT05917041
Title: A Randomised, Open-label, Multicenter, Controlled, Exploratory Study on the Effect and Safety of SAT-001 as a Medical Device in Treatment of Pediatric Patients With Myopia
Brief Title: Exploratory Study of SAT-001 in Treatment of Pediatric Patient With Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT001-KP-001
Record Dates: First submitted 2023-06-12; First posted 2023-06-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-06

CONDITIONS: Children Myopia
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAT-001 (Experimental)
  Interventions: Device: SAT-001(Software as Medical Device)
- Control Group (No Intervention): Wearing glasses or not

INTERVENTIONS:
Device: SAT-001(Software as Medical Device) — Using SAT-001 application for 48 weeks and wearing glasses or not
  Arms: SAT-001

SUMMARY:
The Purpose of this study is to explore the safety and effectiveness of SAT-001, a medical device for the treatment of myopia in pediatric patient with myopia

DETAILED DESCRIPTION:
Myopic pediatric prevalence rate come to increase rapidly globally. This is a clinical trial to explore the safety and effectiveness of SAT-001(as a Software as Medical Device) developed for the treatment of myopia through suppressing the progress myopia

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patient age 5 to 12 years old at the Screening Visit
2. Diagnosed with myopia as following refractive error via cycloplegic refraction(CR)

   1. Spherical equivalent (SE) -0.75 D or more and less than -6.00 D in each eye
   2. Astigmatism of 1.50 D or less in each eye
   3. Anisometropia of less than 1.00 D
3. The age of birth over 38 weeks
4. Over 2500g of birth weight
5. Best corrected distance visual acuity of 0.2 logMAR or better in each eye at the Screening Visit
6. Intraocular pressure 21 mmHg or less in each eye at the Screening Visit

Exclusion Criteria:

1. Administration of anti-muscarine drugs within 1 month before screening visit
2. Current or previous use of multi-focal lenses
3. Planning to use or having used Orthokeratology lenses (Ortho-K lenses), Rigid Gas Permeable (RGP) lenses, and other contact lenses to reduce the progression of myopia
4. History of atropine use for treatment of myopia within 1 month before screening visit
5. Abnormal conditions in cornea, lens, central retina, iris and ciliary bodies or malignant tumors around orbit
6. History of manifest strabismus, intermittent strabismus, amblyopia, nystagmus etc. (except for phoria maintaining binocular vision)
7. History of ophthalmic surgery, such as eyelid surgery, strabismus surgery, intraocular surgery, or refractive correction surgery (except for epiblepharon surgery)
8. Obsessive-compulsive disorder or attention deficit hyperactivity disorder(ADHD)
9. Down's syndrome or cerebral palsy
10. Participation in another clinical trial within 6 months before screening visit
11. History of growth hormone treatment within 1 month before screening visit
12. Medically clear to have abnormal range of intellectual development
13. Significant systemic diseases such as congenital heart disease, respiratory system disease (except for asthma), endocrine disease or nervous system disease
14. Currently taking or having taken antihistamines (tablets, nasal spray, eye drops, etc.) or psychiatric drugs (antidepressants, anti-anxiety medications, etc.) within 30 days before screening visit
15. History of injections with histamine release and cholinergic effect within 30 days before screening visit
16. Incongruent to participate in this study at the discretion of the investigator

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Change in cycloplegic Refraction Error | Baseline, 24 weeks, 48 weeks
Change in axial length | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - HanGil Eye Hospital, Incheon
  - Kangbuk Samsung Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided